CLINICAL TRIAL: NCT03649737
Title: Pilot Study of a Progressive Exercise Program Among Lung Cancer Patient-Partner Dyads
Brief Title: Exercise Program Among Lung Cancer Dyads
Acronym: PEP-LC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Portland VA Medical Center (U.S. Federal Agency); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Donald Sullivan, Assistant Professor, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00018245
Record Dates: First submitted 2018-07-27; First posted 2018-08-28 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Lung Cancer; Depression; Physical Activity; Quality of Life; Pain; Lung Cancer Symptoms
MeSH Terms: conditions — Lung Neoplasms; Depression; Motor Activity; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (exercise) (Experimental): Participants attend supervised group exercises classes twice per week during weeks 1-6 and once per week during weeks 7-12. Participants also attend home-based unsupervised exercise sessions via an instructional DVD once per weeks over for 30 minutes during weeks 1-6 and twice per week during weeks 7-12.
  Interventions: Behavioral: Exercise Intervention; Other: Survey Administration; Other: Quality-of-Life Assessment

INTERVENTIONS:
Behavioral: Exercise Intervention — Attend supervised and unsupervised exercise sessions
Other: Survey Administration — Ancillary studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
Pilot study of an exercise program among patients with all stages of lung cancer examining feasibility and acceptability. Preliminary outcomes include objective measures of physical function, depression, adherence to lung cancer treatments, Quality of Life (QOL), and social support.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the feasibility and acceptability of a progressive exercise program initiated after lung cancer diagnosis among patient partner dyads.

SECONDARY OBJECTIVE:

I. Examine the preliminary effects of partnered exercise on physical function, depression, adherence to lung cancer treatments, QOL and social support .

OUTLINE:

Participants attend supervised group exercises classes twice per week during weeks 1-6 and once per week during weeks 7-12. Participants also attend home-based unsupervised exercise sessions via an instructional DVD once per weeks over for 30 minutes during weeks 1-6 and twice per week during weeks 7-12.

ELIGIBILITY:
Inclusion Criteria:

* Mild depression symptoms
* Able to participate in exercise program per physician approval
* Available partner/spouse to participate with patient

Exclusion Criteria:

* Persistent severe depression symptoms
* Inability to participate in exercise
* Life expectancy less than 1 year

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2019-10-22 (Actual)

PRIMARY OUTCOMES:
Study Feasibility: Proportion enrolled | 12 weeks
  Will be measured as the number of couples who enroll out of those approached. Will evaluate using descriptive statistics.
Study Acceptability: Average attendance | 12 weeks
  Will be measured by the average attendance at sessions over the course of the intervention. This will be calculated as the total number of classes attended divided by the total possible they could have attended over the course of the study. Attendance will be categorized by sessions couples attended together and those where only one partner attends. Will evaluate using descriptive statistics.

SECONDARY OUTCOMES:
Incidence of Depression | 12 weeks
  Will be measured using the Patient Health Questionnaire - 8 (PHQ-8). Total sum scores range from 0-24 with 0 indicating no symptoms to higher scores (>=10) indicating major depressive symptoms.
Change in physical function over time: 6-minute walk | 12 weeks
  We will monitor the change in physical function over time of the participants with lung cancer in our study. Physical functioning will be measured at baseline, week 6, and week 12 of the exercise program. For this test, the participants ability to walk for 6 minutes, and the distance (meters) walked within that 6 minutes will be recorded and compared at each time point.
Change in physical function over time: Hand grip test | 12 weeks
  We will monitor the change in physical function over time of the participants with lung cancer in our study. Physical functioning will be measured at baseline, week 6, and week 12 of the exercise program. For the hand grip test, participants will grip a dynamometer that measures force in kg. The force of the grip will be measured and compared at each time point.
Change in physical function over time: Short Physical Performance Battery | 12 weeks
  We will monitor the change in physical function over time of the participants with lung cancer in our study. Physical functioning will be measured at baseline, week 6, and week 12 of the exercise program. The Short Physical Performance Battery test includes height/weight measurements, standing balance tests (semi-tandem, side-by-side, full tandem), walking speed (at 4 meters), and chair stands. Participants are assigned scores based on their ability to complete each exercise. For the Balance test, 0=incomplete, 1=complete. For the time it takes to walk 4 meters, point values of 1 to 4 are assigned. (1=8.7 sec, 2=6.21 to 8.70 sec, 3=4.82 to 6.20 sec, 4=less than 4.82 sec). For the chair stands, 1=between 16.7 sec and 60 sec, 2=13.7 sec to 16.69 sec, 3=11.2 sec to 13.69 sec, 4=11.19 sec or less. Each of these scores are then summed. The sum scores will be compared at each time point to measure change in physical function over time.
Quality of Life for participants with lung cancer assessed by FACT-L | 12 weeks
  Quality of life for participants with lung cancer will be measured using the Functional Assessment of Cancer Therapy - Lung (FACT-L). The 36-item questionnaire uses a 5-point scale ranging from 0 (Not at all) to 4 (Very Much). We will measure the sum of all responses as well as look at sub-scales: physical, social/family, emotional, functional, and additional concerns.
Quality of Life for exercise partners assessed by CQOLC | 12 weeks
  Quality of life for exercise partners will be measured using the Caregiver Quality of Life Index - Cancer (CQOLC), a 35-item questionnaire about caring for loved ones with lung cancer. It uses a 5-point scale ranging from 0 (Not at all) to 4 (Very much)
Fatigue assessed by PROMIS Short-Form | 12 weeks
  PROMIS® (Patient-Reported Outcomes Measurement Information System) Short-Form - Fatigue questionnaires measure the fatigue experienced in the past 7 days and its level of interference with daily activities. All participants will answer the 7-item questionnaire using a 5-point scale ranging from 0 (Never) to 4 (Always).
Pain assessed by PROMIS Short-Form | 12 weeks
  PROMIS® (Patient-Reported Outcomes Measurement Information System) Short-From - Pain questionnaires measure both pain intensity, quality, and impact on daily function experienced in the past 7 days. All participants will answer the 16 questions using a 5-point Likert scale. Scores range from 0, "no pain" to 4, "very severe"; and 0, "not at all" to 4, "very much."
Sleep assessed by PROMIS Short-Form | 12 weeks
  PROMIS® (Patient-Reported Outcomes Measurement Information System) Short-Form - Sleep questionnaire measures the sleep quality using an 8-item questionnaire on a 5-point scale, with responses ranging from 0 (Very Poor/Not at all) to 4 (Very Good/Not at all).
Relationship Distress assessed by DAS-SF | 12 weeks
  Measured using the DAS-SF (Dyadic Adjustment Scale - Short Form) a 7-item scale asking about relationship satisfaction and scored using a 5-point scale ranging from 1 (Low) to 5 (High)
Social Support assessed by PSSS | 12 weeks
  The Multidimensional Scale of Perceived Social Support (PSSS) is a 12-item questionnaire that uses a 7 point Likert scale that measures the support one receives from friends, family, and significant others.
Level of exercise outside the exercise intervention assessed by GLTEQ | 12 weeks
  The Godin Leisure-Time Exercise Questionnaire (GLTEQ) is a self-report questionnaire asking the patient-participant how often they engaged in mild effort, moderate exercise, strenuous exercise, and resistance (weight bearing exercise). This will be measured in three different ways: 1) total activity = vigorous + moderate + mild + resistance, 2) physical activity guidelines = moderate + (vigorous x 2), 3) moderate + vigorous.
Incidence of Malnutrition | 12 weeks
  Measured using a Malnutrition Screening Tool (MST). Patients with lung cancer with a score of 2 or more are considered at risk for malnutrition.
Subjective evaluation of PEP-LC participant experience from phone interviews | 1-2 months follow completion of program (up to 4 months)
  Dyads participating in the exercise intervention will complete a follow up phone interview regarding their experience in the program. They will be ask to describe their overall experience as well as indicate if they have any suggestions on making the program better
Incidence of Relationship Strain | 12 weeks
  Partner participants will complete the Modified Caregiver Strain Index (MCSI), an 18-item questionnaire about strain caused by caretaking for a person with cancer. Uses a 5-point scale ranging from 0 (Never) to 4 (A great deal)

CONTACTS AND LOCATIONS:
Overall Officials: Donald R Sullivan, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (2):
- United States (2):
  - Oregon Health and Science University, Portland, Oregon
  - VA Portland Health Care System, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Walker J, Holm Hansen C, Martin P, Sawhney A, Thekkumpurath P, Beale C, Symeonides S, Wall L, Murray G, Sharpe M. Prevalence of depression in adults with cancer: a systematic review. Ann Oncol. 2013 Apr;24(4):895-900. doi: 10.1093/annonc/mds575. Epub 2012 Nov 21. PMID 23175625
- [Background] Sullivan DR, Ganzini L, Duckart JP, Lopez-Chavez A, Deffebach ME, Thielke SM, Slatore CG. Treatment receipt and outcomes among lung cancer patients with depression. Clin Oncol (R Coll Radiol). 2014 Jan;26(1):25-31. doi: 10.1016/j.clon.2013.09.001. Epub 2013 Sep 27. PMID 24080122
- [Background] Sullivan DR, Forsberg CW, Ganzini L, Au DH, Gould MK, Provenzale D, Slatore CG. Longitudinal Changes in Depression Symptoms and Survival Among Patients With Lung Cancer: A National Cohort Assessment. J Clin Oncol. 2016 Nov 20;34(33):3984-3991. doi: 10.1200/JCO.2016.66.8459. Epub 2016 Oct 31. PMID 27996350
- [Background] Massie MJ. Prevalence of depression in patients with cancer. J Natl Cancer Inst Monogr. 2004;(32):57-71. doi: 10.1093/jncimonographs/lgh014. PMID 15263042
- [Background] Lyons KS, Miller LM, McCarthy MJ. The Roles of Dyadic Appraisal and Coping in Couples With Lung Cancer. J Fam Nurs. 2016 Nov;22(4):493-514. doi: 10.1177/1074840716675976. Epub 2016 Oct 31. PMID 27803239
- [Background] Brown Johnson CG, Brodsky JL, Cataldo JK. Lung cancer stigma, anxiety, depression, and quality of life. J Psychosoc Oncol. 2014;32(1):59-73. doi: 10.1080/07347332.2013.855963. PMID 24428251
- [Background] Cataldo JK, Jahan TM, Pongquan VL. Lung cancer stigma, depression, and quality of life among ever and never smokers. Eur J Oncol Nurs. 2012 Jul;16(3):264-9. doi: 10.1016/j.ejon.2011.06.008. Epub 2011 Jul 30. PMID 21803653
- [Background] Piderman KM, Sytsma TT, Frost MH, Novotny PJ, Rausch Osian SM, Solberg Nes L, Patten CA, Sloan JA, Rummans TA, Bronars CA, Yang P, Clark MM. Improving Spiritual Well-Being in Patients with Lung Cancers. J Pastoral Care Counsel. 2015 Sep;69(3):156-62. doi: 10.1177/1542305015602711. PMID 26463853
- [Background] Miller LM, Sullivan DR, Lyons KS. Dyadic Perceptions of the Decision Process in Families Living With Lung Cancer. Oncol Nurs Forum. 2017 Jan 1;44(1):108-115. doi: 10.1188/17.ONF.108-115. PMID 27991611
- [Background] Lyons KS, Bennett JA, Nail LM, Fromme EK, Dieckmann N, Sayer AG. The role of patient pain and physical function on depressive symptoms in couples with lung cancer: a longitudinal dyadic analysis. J Fam Psychol. 2014 Oct;28(5):692-700. doi: 10.1037/fam0000017. Epub 2014 Aug 4. PMID 25090253
- [Background] Kim Y, Carver CS, Spillers RL, Crammer C, Zhou ES. Individual and dyadic relations between spiritual well-being and quality of life among cancer survivors and their spousal caregivers. Psychooncology. 2011 Jul;20(7):762-70. doi: 10.1002/pon.1778. Epub 2010 May 25. PMID 20878868
- [Background] Berg CA, Upchurch R. A developmental-contextual model of couples coping with chronic illness across the adult life span. Psychol Bull. 2007 Nov;133(6):920-54. doi: 10.1037/0033-2909.133.6.920. PMID 17967089
- [Background] Brown LF, Kroenke K, Theobald DE, Wu J, Tu W. The association of depression and anxiety with health-related quality of life in cancer patients with depression and/or pain. Psychooncology. 2010 Jul;19(7):734-41. doi: 10.1002/pon.1627. PMID 19777535
- [Background] Lazenby M, Ercolano E, Grant M, Holland JC, Jacobsen PB, McCorkle R. Supporting commission on cancer-mandated psychosocial distress screening with implementation strategies. J Oncol Pract. 2015 May;11(3):e413-20. doi: 10.1200/JOP.2014.002816. Epub 2015 Mar 10. PMID 25758447
- [Background] Walker J, Sawhney A, Hansen CH, Ahmed S, Martin P, Symeonides S, Murray G, Sharpe M. Treatment of depression in adults with cancer: a systematic review of randomized controlled trials. Psychol Med. 2014 Apr;44(5):897-907. doi: 10.1017/S0033291713001372. Epub 2013 Jun 19. PMID 23778105
- [Background] Cooney GM, Dwan K, Greig CA, Lawlor DA, Rimer J, Waugh FR, McMurdo M, Mead GE. Exercise for depression. Cochrane Database Syst Rev. 2013 Sep 12;2013(9):CD004366. doi: 10.1002/14651858.CD004366.pub6. PMID 24026850
- [Background] DiLorenzo TM, Bargman EP, Stucky-Ropp R, Brassington GS, Frensch PA, LaFontaine T. Long-term effects of aerobic exercise on psychological outcomes. Prev Med. 1999 Jan;28(1):75-85. doi: 10.1006/pmed.1998.0385. PMID 9973590
- [Background] Buffart LM, Kalter J, Sweegers MG, Courneya KS, Newton RU, Aaronson NK, Jacobsen PB, May AM, Galvao DA, Chinapaw MJ, Steindorf K, Irwin ML, Stuiver MM, Hayes S, Griffith KA, Lucia A, Mesters I, van Weert E, Knoop H, Goedendorp MM, Mutrie N, Daley AJ, McConnachie A, Bohus M, Thorsen L, Schulz KH, Short CE, James EL, Plotnikoff RC, Arbane G, Schmidt ME, Potthoff K, van Beurden M, Oldenburg HS, Sonke GS, van Harten WH, Garrod R, Schmitz KH, Winters-Stone KM, Velthuis MJ, Taaffe DR, van Mechelen W, Kersten MJ, Nollet F, Wenzel J, Wiskemann J, Verdonck-de Leeuw IM, Brug J. Effects and moderators of exercise on quality of life and physical function in patients with cancer: An individual patient data meta-analysis of 34 RCTs. Cancer Treat Rev. 2017 Jan;52:91-104. doi: 10.1016/j.ctrv.2016.11.010. Epub 2016 Dec 5. PMID 28006694
- [Background] Speck RM, Courneya KS, Masse LC, Duval S, Schmitz KH. An update of controlled physical activity trials in cancer survivors: a systematic review and meta-analysis. J Cancer Surviv. 2010 Jun;4(2):87-100. doi: 10.1007/s11764-009-0110-5. Epub 2010 Jan 6. PMID 20052559
- [Background] Cavalheri V, Jenkins S, Cecins N, Gain K, Phillips MJ, Sanders LH, Hill K. Exercise training for people following curative intent treatment for non-small cell lung cancer: a randomized controlled trial. Braz J Phys Ther. 2017 Jan-Feb;21(1):58-68. doi: 10.1016/j.bjpt.2016.12.005. Epub 2017 Jan 13. PMID 28442076
- [Background] Cavalheri V, Tahirah F, Nonoyama M, Jenkins S, Hill K. Exercise training undertaken by people within 12 months of lung resection for non-small cell lung cancer. Cochrane Database Syst Rev. 2013 Jul 31;(7):CD009955. doi: 10.1002/14651858.CD009955.pub2. PMID 23904353
- [Background] Winters-Stone KM, Moe EL, Perry CK, Medysky M, Pommier R, Vetto J, Naik A. Enhancing an oncologist's recommendation to exercise to manage fatigue levels in breast cancer patients: a randomized controlled trial. Support Care Cancer. 2018 Mar;26(3):905-912. doi: 10.1007/s00520-017-3909-z. Epub 2017 Sep 30. PMID 28965138
- [Background] Winters-Stone KM, Li F, Horak F, Luoh SW, Bennett JA, Nail L, Dieckmann N. Comparison of tai chi vs. strength training for fall prevention among female cancer survivors: study protocol for the GET FIT trial. BMC Cancer. 2012 Dec 5;12:577. doi: 10.1186/1471-2407-12-577. PMID 23217054
- [Background] Winters-Stone KM, Lyons KS, Dobek J, Dieckmann NF, Bennett JA, Nail L, Beer TM. Benefits of partnered strength training for prostate cancer survivors and spouses: results from a randomized controlled trial of the Exercising Together project. J Cancer Surviv. 2016 Aug;10(4):633-44. doi: 10.1007/s11764-015-0509-0. Epub 2015 Dec 29. PMID 26715587
- [Background] Kamen C, Heckler C, Janelsins MC, Peppone LJ, McMahon JM, Morrow GR, Bowen D, Mustian K. A Dyadic Exercise Intervention to Reduce Psychological Distress Among Lesbian, Gay, and Heterosexual Cancer Survivors. LGBT Health. 2016 Feb;3(1):57-64. doi: 10.1089/lgbt.2015.0101. Epub 2015 Nov 24. PMID 26652029
- [Background] Rasekaba T, Lee AL, Naughton MT, Williams TJ, Holland AE. The six-minute walk test: a useful metric for the cardiopulmonary patient. Intern Med J. 2009 Aug;39(8):495-501. doi: 10.1111/j.1445-5994.2008.01880.x. PMID 19732197
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Andersen BL, Rowland JH, Somerfield MR. Screening, assessment, and care of anxiety and depressive symptoms in adults with cancer: an american society of clinical oncology guideline adaptation. J Oncol Pract. 2015 Mar;11(2):133-4. doi: 10.1200/JOP.2014.002311. Epub 2014 Dec 16. No abstract available. PMID 25515721
- [Background] Zimet GD, Powell SS, Farley GK, Werkman S, Berkoff KA. Psychometric characteristics of the Multidimensional Scale of Perceived Social Support. J Pers Assess. 1990 Winter;55(3-4):610-7. doi: 10.1080/00223891.1990.9674095. PMID 2280326
- [Background] Wright SP, Hall Brown TS, Collier SR, Sandberg K. How consumer physical activity monitors could transform human physiology research. Am J Physiol Regul Integr Comp Physiol. 2017 Mar 1;312(3):R358-R367. doi: 10.1152/ajpregu.00349.2016. Epub 2017 Jan 4. PMID 28052867
- [Background] Zhang X, McClean D, Ko E, Morgan MA, Schmitz K. Exercise Among Women With Ovarian Cancer: A Feasibility and Pre-/Post-Test Exploratory Pilot Study. Oncol Nurs Forum. 2017 May 1;44(3):366-374. doi: 10.1188/17.ONF.366-374. PMID 28635971
- [Background] Guralnik JM, Ferrucci L, Simonsick EM, Salive ME, Wallace RB. Lower-extremity function in persons over the age of 70 years as a predictor of subsequent disability. N Engl J Med. 1995 Mar 2;332(9):556-61. doi: 10.1056/NEJM199503023320902. PMID 7838189
- [Background] Newman AB, Simonsick EM, Naydeck BL, Boudreau RM, Kritchevsky SB, Nevitt MC, Pahor M, Satterfield S, Brach JS, Studenski SA, Harris TB. Association of long-distance corridor walk performance with mortality, cardiovascular disease, mobility limitation, and disability. JAMA. 2006 May 3;295(17):2018-26. doi: 10.1001/jama.295.17.2018. PMID 16670410
- [Background] Eickmeyer SM, Walczak CK, Myers KB, Lindstrom DR, Layde P, Campbell BH. Quality of life, shoulder range of motion, and spinal accessory nerve status in 5-year survivors of head and neck cancer. PM R. 2014 Dec;6(12):1073-80. doi: 10.1016/j.pmrj.2014.05.015. Epub 2014 May 28. PMID 24880060
- [Background] Stark T, Walker B, Phillips JK, Fejer R, Beck R. Hand-held dynamometry correlation with the gold standard isokinetic dynamometry: a systematic review. PM R. 2011 May;3(5):472-9. doi: 10.1016/j.pmrj.2010.10.025. PMID 21570036
- [Background] Ameringer S, Elswick RK Jr, Menzies V, Robins JL, Starkweather A, Walter J, Gentry AE, Jallo N. Psychometric Evaluation of the Patient-Reported Outcomes Measurement Information System Fatigue-Short Form Across Diverse Populations. Nurs Res. 2016 Jul-Aug;65(4):279-89. doi: 10.1097/NNR.0000000000000162. PMID 27362514
- [Derived] Leng QL, Lyons KS, Winters-Stone KM, Medysky ME, Dieckmann NF, Denfeld QE, Sullivan DR. Preliminary effects of a yoga intervention for lung cancer dyads: benefits for care partners. Support Care Cancer. 2024 Jun 20;32(7):447. doi: 10.1007/s00520-024-08638-5. PMID 38902487